CLINICAL TRIAL: NCT05102370
Title: A Pilot Study of Enasidenib for Patients With Clonal Cytopenia of Undetermined Significance and Mutations in IDH2
Brief Title: A Study of Enasidenib in People With Clonal Cytopenia of Undetermined Significance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-268
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Clonal Cytopenia of Undetermined Significance; CCUS Clonal Cytopenia of Undetermined Significance
Keywords: CCUS; Clonal Cytopenia of Undetermined Significance; Enasidenib; 21-268; Memorial Sloan Kettering Cancer Center
MeSH Terms: interventions — enasidenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with CCUS with mutations in IDH2 (Experimental): Participants will have CCUS with mutations in IDH2
  Interventions: Drug: Enasidenib

INTERVENTIONS:
Drug: Enasidenib — Study participants will receive enasidenib 100 mg daily for 18 months. Participants will continue treatment with enasidenib until confirmed progression to AML or MDS, development of unacceptable toxicity, or suspicion of disease progression, provided the patient is deriving clinical benefit, which will be determined at the discretion of the principal investigator.

SUMMARY:
Study researchers think that a drug called enasidenib may help people with clonal cytopenia of undetermined significance (CCUS) because the drug blocks the mutated IDH2 protein, which may improve blood cell counts. The purpose of this study is to find out whether enasidenib is a safe and effective treatment for CCUS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of signing the informed consent form.
* Willing and able to adhere to the study visit schedule and other protocol requirements.
* Unexplained cytopenia for at least 6 months. Cytopenia is defined as the presence of ≥1 blood count indexes below the following thresholds:
* Hgb <10 g/dL
* ANC <1.8 × 10^9/L
* Platelets <100 × 10^9/L
* Results of bone marrow biopsy within 1 month of study entry (screening bone marrow biopsy) must not indicate hematologic disease.
* IDH2 gene mutation (R140 or R172), performed locally, at a frequency >2%.
* ECOG performance status of 0-2.
* Adequate organ function, defined as:

  * Serum aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤3x upper limit of normal (ULN), unless the subject has Gilbert's syndrome.
  * Serum total bilirubin <1.5x ULN. Higher levels are acceptable if these can be attributed to ineffective erythropoiesis. In these cases, approval from the study Principal Investigator is required.
  * Creatinine clearance greater than 50 mL/min based on the Cockroft-Gault glomerular filtration rate estimation.
* Patients being enrolled on study on the basis of anemia, will only be eligible if folate, B12, serum iron, serum ferritin, total iron binding capacity, haptoglobin and peripheral smear within normal limits
* Women of childbearing potential may participate provided they have a negative serum pregnancy test at screening and a negative serum or urine pregnancy test within 72 h of starting treatment.
* Women of childbearing potential (WOCBP) and males with partners who are WOCBP must agree to abstain from sexual intercourse or to use 1 highly effective form of contraception during the study and for at least 4 months following the last dose of enasidenib. Males with partners who are WOCBP must agree to use a barrier method.

Exclusion Criteria:

* Active malignancy defined as >1-cm disease on most recent CT scan in the past 6 months or recent history of cancer (i.e. within the past 5 years) with >50% chance of cancer recurrence in the next 5 years.
* Current or prior history of hematologic malignancy.
* Therapy (including maintenance therapy) for solid-tumor malignancy within the last 6 months.
* Known dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.
* Active uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment).
* Positive direct Coombs test
* Evidence of hypersplenism on physical exam
* Pregnant or lactating (women).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2026-01-26 (Actual); Study Completion 2026-01-26 (Actual)

PRIMARY OUTCOMES:
Best Response | Up to 18 months
  The primary objective is to estimate the rate of hematologic improvement. The endpoint is evaluated as the best response at any point in up to 18 months of treatment with enasidenib.

CONTACTS AND LOCATIONS:
Overall Officials: Eytan Stein, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (12):
- United States (12):
  - Mayo Clinic (Data Collection Only), Rochester, Minnesota
  - Washington University (Data Collection and Specimen Analysis), St Louis, Missouri
  - Memorial Sloan Kettering at Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Rockville Centre, New York
  - Cleveland Clinic (Data Collection Only), Cleveland, Ohio
  - Ohio State University (Data Collection Only), Columbus, Ohio
  - Oregon Health & Science University (Data Collection Only), Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org